CLINICAL TRIAL: NCT07359573
Title: Evaluating and Monitoring Physical Fatigue While Performing Functional Activities
Brief Title: The Effect of a Passive Hip Exoskeleton on Daily-life Fatigue in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, David Beckwee, Associate Professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RevalExo_Exoband
Record Dates: First submitted 2025-12-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fatigue; Older Adults (65 Years and Older)
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exoband ON (Active Comparator): The participants execute the fatigue protocol while wearing the passive hip exoskeletons (Exoband).
  Interventions: Other: Performance test; Device: Exoband
- Exoband OFF (Placebo Comparator): The participants execute the fatigue protocol without wearing the passive hip exoskeletons (Exoband).
  Interventions: Other: Performance test

INTERVENTIONS:
Other: Performance test — The participant will be asked to execute a protocol in the movement lab that induces progressive feelings of fatigue. This protocol includes a sequence of relevant functional activities, such as stair walking, slope walking, crouching, walking different path shapes. During this execution the Ratings of Perceived Exertion will be questioned, and simultaneously physiological and movement data will be collected.
Device: Exoband — The participant will wear the Exoband (Moveo), which is a lightweight, soft wearable exoskeleton designed to assist walking by providing elastic support to the hip during gait. It uses passive elastic elements to store and release energy in sync with the user's movement, reducing muscular effort without motors or batteries. The system is unobtrusive and aims to support mobility while preserving natural movement patterns.
  Arms: Exoband ON

SUMMARY:
This crossover study investigates whether a passive lower-limb exoskeleton (Exoband) can reduce perceived exertion during everyday mobility tasks in older adults. Participants complete the fatigue protocol- a structured sequence of daily challenging tasks (e.g., overground walking, stair and slope walking, obstacle avoidance)-once with the Exoband and once without it, in randomized order and separated by a one-week washout period. During each session, distance covered until fatigue, rate of perceived exertion, physiological and gait parameters are recorded. The aim is to determine whether exoskeleton assistance enhances mobility performance and reduces functional fatigue across older adults.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old
* Healthy physical condition

Exclusion Criteria:

* Physical injury or disorder that doesn't allow good physical performance

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the Ratings of Perceived Exertion throughout the protocol execution | Through study completion, an average of 1-2 weeks.
  The subjective feelings of fatigue will be evaluated through the Ratings of Perceived Exertion, using the modified Borg Scale (score ranging from 0 'no exertion' to 10 'maximal exertion'). This will be expressed verbally by the participant throughout the execution of the protocol.

SECONDARY OUTCOMES:
Changes in muscle activity (surface EMG) throughout the protocol execution | Through study completion, an average of 1-2 weeks.
  Muscle activity data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in heart rate (variability) (ECG sensors) throughout the protocol execution | Through study completion, an average of 1-2 weeks.
  Cardiorespiratory data (Heart rate) will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in muscle oxygen saturation (Moxy Monitor) throughout the protocol execution | Through study completion, an average of 1-2 weeks.
  Oxygen saturation data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in electrodermal activity (Galvanic Skin Response - finger electrodes) throughout the protocol execution | Through study completion, an average of 1-2 weeks.
  Electrodermal activity data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in motion data (IMU sensors) throughout the protocol execution | Through study completion, an average of 1-2 weeks.
  Inertial Measurement Unit (IMU) data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in respiratory rate (respiratory chest band) throughout the protocol execution | Through study completion, an average of 1-2 weeks.
  Respiratory data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.

CONTACTS AND LOCATIONS:
Overall Officials: David Beckwée, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Brubotics Rehabilitation Research Center, Jette, Brussels Capital, Belgium